CLINICAL TRIAL: NCT06326411
Title: A Phase I, Open Label Single-arm Two-part Study to Investigate Safety, Pharmacokinetics, and Preliminary Efficacy of Pan-RAF/MEK Glue NST-628 Oral Tablets in Subject With Solid Tumors Harboring Genetic Alterations in the MAPK Pathway and With Other Solid Tumors
Brief Title: A Study to Investigate the Safety and Efficacy of NST-628 Oral Tablets in Subjects With Solid Tumors
Acronym: NST-628
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nested Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NST-628-001
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-06

CONDITIONS: Oncology; MEK Mutation; RAF Gene Mutation; Ras (KRAS or NRAS) Gene Mutation; Melanoma; NSCLC; Glioma; Solid Tumor, Adult; MAPK Pathway Gene Mutation
Keywords: RAS; MEK; RAF; solid tumor
MeSH Terms: conditions — Neoplasms; Melanoma; Glioma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part A Dose Escalation and Part B Dose Expansion (Experimental): Part A will evaluate the safety of NST-628 with advanced solid tumors and determine the recommended dose for expansion of NST-628.
  Part B will evaluate the objective tumor response rate in subjects with advanced solid tumors harboring specified genetic alterations receiving NST-628 and evaluate the safety of NST-628 in subjects with advanced solid tumors in cohorts defined below:
  i. Melanoma Cohorts
  1. Activating NRAS mutations
  2. Select BRAF alterations
  ii. Non-Melanoma Cohorts:
  1. Solid tumors with NRAS activating mutations
  2. Solid tumors with KRAS activating mutations
  3. Solid tumors with select BRAF alterations
  4. Glioma with BRAF alterations
  Interventions: Drug: NST-628

INTERVENTIONS:
Drug: NST-628 — NST-628 is a small molecule non-covalent pan-RAF/MEK dual molecular glue targeting RAF and MEK nodes of MAPK pathway.

SUMMARY:
This is a two-part Phase 1, open label, multi-center, single arm, non-randomized, multiple dose, safety, pharmacokinetic (PK) and preliminary efficacy study of single agent NST-628 in adult patients with MAPK pathway mutated/dependent advanced solid tumors who have exhausted standard treatment options.

DETAILED DESCRIPTION:
The study includes two parts, a dose escalation part (Part A) followed by a dose expansion part (Part B). Part A will estimate the maximum tolerated dose (MTD) in dose escalation cohorts in patients with advanced solid tumors for whom no standard therapy is available in order to establish the recommended dose for expansion (RDE). Successive cohorts of subjects will receive escalating doses of NST-628 orally once daily in 28-day cycles.

Bayesian Optimal Interval (BOIN) method will be used for dose escalation.

Once MTD is reached or dose escalation is stopped prior to reaching MTD and provisional RDE selected, the provisional RDE level will be expanded. If warranted by dose/toxicity/anti-tumor activity observations, additional, lower dose level(s) may also be expanded.

Part B of the study will include up to 6 cohorts of approximately up to 30 subjects each with select MAPK pathway mutant solid tumors enrolled at the RDE in order to explore benefit from treatment as suggested by preclinical findings and will better define the safety profile of NST-628 at the RDE. Additional safety information gathered in Part B may be used to modify the dose recommended for future studies.

The end of the study is the last visit of the last subject.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible to be included in the study only if all of the following criteria apply:

1. Subjects must be ≥18 years old (or of legal age of consent in the country in which the study is taking place) at the time of signing the informed consent.
2. Subjects who have a histologically or cytologically documented metastatic or locally advanced solid tumor, for which standard of care (SoC) therapy does not exist, no longer provides benefit, or is not tolerated by the subject, or the subject has been assessed by the Investigator as not being suitable for SoC therapy.

   1. Part A: Subjects with any solid tumor with genetic alteration of or evidence of tumor dependence upon the RAS/MAPK pathway (subject to additional restrictions specified in the study protocol)
   2. Part B: Subjects must be diagnosed with one of the following solid tumors harboring specified genetic alterations based on a validated local test:

   i. Melanoma Cohorts:
   1. Activating NRAS mutations
   2. Select BRAF alterations

   ii. Non-Melanoma Cohorts:
   1. Solid tumors with NRAS activating mutations
   2. Solid tumors with KRAS activating mutations
   3. Solid tumors with select BRAF alterations
   4. Glioma with BRAF alterations
3. Newly obtained or archived tumor tissue is required
4. Part B: measurable disease as defined by RECIST Version 1.1 or by other disease assessment tool standard for a given tumor type (if RECIST v. 1.1 is not standard)
5. Performance status

   1. Solid tumors other than glioma: ECOG 0 or 1
   2. Glioma: Karnofsky ≥ 70 and ECOG 0 or 1
6. Have adequate organ function
7. Understand and voluntarily sign an Institutional Review Board/Independent Ethics Committee-approved informed consent form prior to any study-specific evaluation.
8. Life expectancy ≥ 12 weeks

Exclusion Criteria:

Subjects are excluded from the study if any of the following criteria apply:

1. Conditions interfering with oral intake of NST-628
2. Conditions interfering with intestinal absorption of an orally administered drug
3. A history or current evidence of significant retinal pathology leading to increased risk of RVO
4. A history or evidence of cardiovascular risk
5. Current or history within 6 months of planned Cycle 1 Day 1 of pneumonitis or interstitial lung disease (ILD)
6. Part B: prior treatment with any MEK or BRAF inhibitor
7. Untreated or symptomatic central nervous system (CNS) metastases
8. Chemotherapy, radiation, gene therapy, vaccine therapy, or anti-cancer antibodies / ADCs within 28 days of Cycle 1 Day 1
9. Targeted small molecule agents within 14 days or 5 half-lives of Cycle 1 Day 1
10. Females who are pregnant or breastfeeding.
11. For fertile patients (female able to become pregnant or male able to father a child), refusal to use effective contraception during the period of the trial and for 6 months after the last dose of NST-628
12. Presence of any serious or unstable concomitant systemic disorder incompatible with the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Part A and B: Evaluate the safety of NST-628 in patients with advanced solid tumors | Through study completion, an average of 1 year
  Adverse effects
Part A: Determine the recommended dose for expansion of NST-628 | The first 28 days of treatment (DLTs)
  Dose limiting toxicities (DLTs)
Part B: Evaluate objective tumor response rate | Through study completion, an average of 1 year
  Objective response per RECIST v. 1.1 or other response assessment tool standard for a given tumor type.

SECONDARY OUTCOMES:
Part A: Evaluate objective tumor response rate | Through study completion, an average of 1 year
  Objective response per RECIST v. 1.1 or other response assessment tool standard for a given tumor type.
Part A and B: Evaluate progression free survival (PFS) | Through study completion, an average of 1 year
  PFS defined as the time to first occurrence of disease progression per RECIST v1.1 (or other response assessment tool standard for a given tumor type) or death
Part A and B: Evaluate overall survival (OS) | Through study completion, an average of 2 years
  Overall survival (OS) defined as the time to death
Part A and B: Characterize the pharmacokinetics of NST-628 | Through study completion, an average of 1 year
  NST-628 concentrations in plasma

CONTACTS AND LOCATIONS:
Locations (23):
- United States (17):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - UCLA Hematology/Oncology, Westwood, Los Angeles, California
  - Sarah Cannon Research Institute at Health ONE, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Roswell Park, Buffalo, New York
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Slone Kettering Cancer Center, New York, New York
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - SCRI Oncology Partners, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - NEXT Oncology - Austin, Austin, Texas
  - NEXT Oncology - Dallas, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - START Moutain Region, West Valley City, Utah
  - NEXT Oncology - Virginia, Fairfax, Virginia
- Australia (6):
  - The Kinghorn Cancer Center, St. Vincent's Health Network, Darlinghurst, New South Wales
  - Scientia Clinical Research, Ltd, Randwick, New South Wales
  - Gallipoli Medical Research Centre- Greenslopes Private Hospital, Greenslopes, Queensland
  - Southern Oncology Research Unit, Adelaide, South Australia
  - Cabrini Health Limited, Malvern, Victoria
  - Cabrini Hospital, Malvern, Victoria

IPD SHARING:
Plan to Share IPD: No